CLINICAL TRIAL: NCT03689257
Title: Prospective and Multicenter Study About the Epidemiology and the Characteristics "Omics" in Patients Recently Diagnosed of Inflammatory Bowel Disease in Spain
Brief Title: Study to Evaluate the Epidemiology and the Characteristics "Omics" in Patients Recently Diagnosed of Inflammatory Bowel Disease in Spain
Acronym: IBDomics
Status: Completed | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Responsible Party: Sponsor
Other Study IDs: GIS-2016-IBDomics
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: inflammatory bowel disease; Ulcerative colitis; Crohn´s disease; epidemiology; incidence; omics
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of blood, urine simple and stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective, observational, multicenter, population-based incidence cohort study which will enroll cases of inflammatory bowel disease IBD (Crohn´s disease CD, ulcerative colitis UC, or indeterminate colitis) diagnosed in adults over 18 months in Spain.

In addition, each incident case that gave his/her informed consent, will be followed up for 12 months to determine changes in phenotype or disease location, the need for immunosuppressive and biologic treatments, and the need for hospital admissions and surgery during the first year after diagnosis.

Also, samples of of blood, urine and stool will be collected during the first year after diagnosis

DETAILED DESCRIPTION:
STUDY DESIGN This is a prospective, observational, multicenter, population-based incidence cohort study which will enroll cases of IBD (CD, UC, or indeterminate colitis) diagnosed in adults over 18 months in Spain.

In addition, each incident case that gave his/her informed consent, will be followed up for 12 months to determine changes in phenotype or disease location, the need for immunosuppressive and biologic treatments, and the need for hospital admissions and surgery during the first year after diagnosis.

Samples of blood, urine and stool will be collected during the study visits.

To achieve the aims this study will be Split in two studies.

1. Epidemiology study to achieve aims 1 and 2.
2. Characterization "omics" study to achieve aims 3, 4 and 5.

CASES DETECION

Case detection In Spain, health care is performed mostly by the public health services. According to recent data, approximately 15% of the Spanish population has private health insurance (Informe Sanidad Privada: Aportando Valor. Análisis de situación 2014 (Report on Private Health Care: Providing Value. 2014 Situation Analysis); available at: https://www.fundacionidis.com/wp-content/informes/informe_analisis situac_2014_0.pdf). In addition, of those persons having private health insurance, only about 15% make exclusive use of it. For these reasons and taking into account the specific characteristics of IBD, the risk of underestimating the incidence of IBD considering only cases seen in public health centers would be of little relevance. Therefore, this study will be conducted at centers providing public health care within the National Health System.

To conduct this research project, an IBD specialist who is a member of GETECCU has been selected from each Autonomous Community, who will include patients from their health area.

Each participating investigator will confirm the diagnosis at the time of entering patients in the study and 3 months later to assure this diagnosis and the phenotypic characteristics of the disease, and thereby have greater diagnostic accuracy. External monitoring of incident cases included in the registry will also be performed by review of cases selected at random by the research team of Hospital Universitario de la Princesa.

DEFINITIONS

* Disease location and phenotype: IBD location and phenotype will be defined according to the Montreal classification.
* Time to diagnosis: It will be defined as the time from the first medical consultation made by the patient after onset of symptoms to the diagnosis of IBD.
* Population center: The type of population center at the patient's birth and at diagnosis of IBD will be recorded. Whether the population center of origin of the patient is considered rural or urban will be based on the classification of the National Statistics Institute (INE) of each municipality.
* Socioeconomic level: Socioeconomic level will be assessed through different variables, such as the patient's educational level (primary education or lower, secondary education, higher education or equivalent), occupational status (self-employed, employee, unemployed, retired), professional status (nonsalaried or salaried) and type of working hours (full time or part time).
* Number of cohabitants: The number of cohabitants in the patient's home during childhood (up to 16 years) and at diagnosis of IBD will be recorded.
* Smoking: Smoking status will be categorized as "nonsmoker", "smoker", or "ex-smoker", and will be considered at the time of diagnosis of IBD. Patients will be considered "smokers" if they have a smoked more than 7 cigarettes per week for at least 6 months or smoked at least 1 cigarette in the 6 months prior to diagnosis. Patients will be considered "ex-smokers" l if they quit smoking at least 6 months before diagnosis. Patients will be considered "nonsmokers" if they never smoked or did so in a very small amount or occasionally.
* Treatments: Treatments received by the patient in the 12 months since diagnosis of the disease will be included, provided they were received for IBD. Only the first prescription of each therapeutic group will be recorded.
* Changes in phenotype: Changes in phenotype will be considered as the appearance of new lesions not present at diagnosis subsequent to the initial tests performed to determine disease extent and severity. In these cases, the phenotype, the complication leading to classification of the patient in a different phenotype and date of occurrence of the complication will be recorded.
* Hospital admission Hospital admission occurring during the first year from diagnosis of the disease will be included. The date of admission, date of discharge, if related or not to IBD and the cause of admission.
* Surgical procedures: The surgical procedures performed on the patient since diagnosis of IBD (including those performed before knowing the patient had IBD and which led to its diagnosis), the indication for surgery and the date of surgery will be recorded. An emergency surgical procedure will be considered as any surgery performed within 24 from admission of the patient to the emergency department. An elective surgical procedure will be considered as any procedure performed subsequent to the first day of admission and by the usual surgical team.

DATA COLLECTION

Epidemiology study:

Demographic data (age, sex, smoking), family history of IBD, socioeconomic characteristics, IBD type, pattern, and location and presence of extraintestinal manifestations at diagnosis will collected from each patient. The occurrence of complications (fistulas, stenosis, abscesses), changes in disease location, treatments for IBD, surgeries for IBD, and hospital admission during the first year since diagnosis will also be recorded.

Characterization "omics" study Samples of blood, urine and stool. Date of collection and number of samples.

STUDY VISITS

* Visit 0 (baseline): inclusion of patient in the study and collection of socioeconomic data and on diagnosis of IBD. Collection samples of blood, urine and stool.
* Visit 1 (month 3): confirmation of IBD diagnosis and updating of data related to treatment, changes in phenotype, hospital admissions, and surgery. Collection samples of blood, urine and stool.
* Visit 2 (month 12): confirmation of IBD diagnosis and updating of data related to treatment, changes in phenotype, hospital admissions, and surgery. Collection samples of blood, urine and stool. End of study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age diagnosed of inflammatory bowel disease
* Diagnosis of IBD according to European Crohns and Colitis Organisation (ECCO) criteria.
* The patient must belong to the health area of one of the participating center
* Patients who have accepted to participate in the epidemiology study
* < 1 month since the date of the diagnosis colonoscopy

Exclusion Criteria:

* Patients who do not belong to the health area of the participating centers
* Patients who do not accept to participate in the study
* Patients who have initiated a treatment to IBD
* Patients who received a immunomodulators to treat other disease
* Patients with a immune-mediates systemic disease
* Patients with a active infection or a malignancy in the baseline
* Pregnant patients or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recently diagnosed of inflammatory bowel disese who have not initiated a treatment to IBD
Sampling Method: Non-Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Incidence of IBD in Spain | 1 year
  Measure the incidence of IBD in Spain

SECONDARY OUTCOMES:
Characteristics of patients at diagnosis of inflammatory bowel disease and resources used in the first year after diagnosis | 1 year
  Type of IBD, extension of the IBD, severity of the IBD at diagnosis. Immunosuppressive treatments, biologic drugs, surgery, and hospital
Create a wide collection of samples | 1 year
  Blood simple, urine simple, stool sample
Identify the molecular and cellular pathways involved with IBD development and pathogenesis. | 1 year
  To describe the serum proteomic profile and to characterize the density and composition of serum extracellular vesicles in newly diagnosed IBD patients, aiming to identify the molecular and cellular pathways involved with IBD development and pathogenesis.
Correlate the serum proteomic profile and the density | 1 year
  To correlate the serum proteomic profile and the density and composition of serum extracellular vesicles with IBD phenotype at diagnose and its subsequent evolution during the first year.

CONTACTS AND LOCATIONS:
Locations (16):
- Spain (16):
  - Hospital Universitario Mutua Terrasa, Terrassa, Barcelona
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Santiago de Compostela, Santiago de Compostela, Santiago de Comostela
  - Hospital de Galdakao, Galdakao, Vizcaya
  - Hospital General universitario de Alicante, Alicante
  - Hospital Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital San Jorge, Huesca
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Morale Mesenguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Hospital Universitaro Marqués de Valdecilla, Santander
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Univesitario de Valladolid, Valladolid

REFERENCES:
- [Background] M'Koma AE. Diagnosis of inflammatory bowel disease: Potential role of molecular biometrics. World J Gastrointest Surg. 2014 Nov 27;6(11):208-19. doi: 10.4240/wjgs.v6.i11.208. PMID 25429322
- [Background] M'Koma AE. Inflammatory bowel disease: an expanding global health problem. Clin Med Insights Gastroenterol. 2013 Aug 14;6:33-47. doi: 10.4137/CGast.S12731. eCollection 2013. PMID 24833941
- [Background] Loftus EV Jr. Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences. Gastroenterology. 2004 May;126(6):1504-17. doi: 10.1053/j.gastro.2004.01.063. PMID 15168363
- [Background] Vegh Z, Burisch J, Pedersen N, Kaimakliotis I, Duricova D, Bortlik M, Avnstrom S, Vinding KK, Olsen J, Nielsen KR, Katsanos KH, Tsianos EV, Lakatos L, Schwartz D, Odes S, Lupinacci G, De Padova A, Jonaitis L, Kupcinskas L, Turcan S, Tighineanu O, Mihu I, Barros LF, Magro F, Lazar D, Goldis A, Fernandez A, Hernandez V, Niewiadomski O, Bell S, Langholz E, Munkholm P, Lakatos PL; EpiCom-group. Incidence and initial disease course of inflammatory bowel diseases in 2011 in Europe and Australia: results of the 2011 ECCO-EpiCom inception cohort. J Crohns Colitis. 2014 Nov;8(11):1506-15. doi: 10.1016/j.crohns.2014.06.004. Epub 2014 Jul 4. PMID 24998983
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Fernandez A, Hernandez V, Martinez-Ares D, Sanroman L, de Castro ML, Pineda JR, Carmona A, Gonzalez-Portela C, Salgado C, Martinez-Cadilla J, Pereira S, Garcia-Burriel JI, Vazquez S, Rodriguez-Prada I; EpiCom Group. Incidence and phenotype at diagnosis of inflammatory bowel disease. Results in Spain of the EpiCom study. Gastroenterol Hepatol. 2015 Nov;38(9):534-40. doi: 10.1016/j.gastrohep.2015.03.001. Epub 2015 Apr 15. PMID 25890448
- [Background] Lucendo AJ, Hervias D, Roncero O, Lorente R, Bouhmidi A, Angueira T, Verdejo C, Saluena I, Gonzalez-Castillo S, Arias A. Epidemiology and temporal trends (2000-2012) of inflammatory bowel disease in adult patients in a central region of Spain. Eur J Gastroenterol Hepatol. 2014 Dec;26(12):1399-407. doi: 10.1097/MEG.0000000000000226. PMID 25341061
- [Background] Anton Martinez J, Ortega Gomez A, Arranz Carrero A, Molina Sanchez A, Alvarez Garcia JF, Moreiras Jimenez JL, Gonzalez Blanco P, Gutierrez Sampedro N, Torres Garcia E. [Incidence of inflammatory bowel disease in the health area of Navalmoral de la Mata (Caceres, Spain) between 2000 and 2009]. Gastroenterol Hepatol. 2010 Dec;33(10):694-9. doi: 10.1016/j.gastrohep.2010.08.004. Epub 2010 Nov 3. Spanish. PMID 21051113
- [Background] Lopez-Serrano P, Perez-Calle JL, Carrera-Alonso E, Perez-Fernandez T, Rodriguez-Caravaca G, Boixeda-de-Miguel D, Fernandez-Rodriguez CM. Epidemiologic study on the current incidence of inflammatory bowel disease in Madrid. Rev Esp Enferm Dig. 2009 Nov;101(11):768-72. doi: 10.4321/s1130-01082009001100004. PMID 20001154
- [Background] Arin Letamendia A, Burusco Paternain MJ, Borda Celaya F, Pueyo Royo A, Martinez Echeverria A, Jimenez Perez FJ. Epidemiological aspects of inflammatory bowel disease in the Pamplona area. Rev Esp Enferm Dig. 1999 Nov;91(11):769-76. English, Spanish. PMID 10601770
- [Background] Garrido A, Martinez MJ, Ortega JA, Lobato A, Rodriguez MJ, Guerrero FJ. Epidemiology of chronic inflammatory bowel disease in the Northern area of Huelva. Rev Esp Enferm Dig. 2004 Oct;96(10):687-91; 691-4. doi: 10.4321/s1130-01082004001000003. English, Spanish. PMID 15537375
- [Background] Saro Gismera C, Lacort Fernandez M, Arguelles Fernandez G, Anton Magarzo J, Garcia Lopez R, Navascues CA, Suarez Gonzalez A, Diaz Alvarez G, Gonzalez Bernal A, Palacios Galan A, Altadill Arregui A, Vizoso F. [Incidence and prevalence of inflammatory bowel disease in Gijon, Asturias, Spain]. Gastroenterol Hepatol. 2000 Aug-Sep;23(7):322-7. Spanish. PMID 11002532
- [Background] Monferrer Guardiola R, Martin Jimenez JA, Pedraza Sanz RG, Moreno Sanchez I, Soler Bahilo E, Hinojosa del Val J. Incidence of inflammatory bowel disease in the 02 health area of Castellon (1992-1996). Rev Esp Enferm Dig. 1999 Jan;91(1):33-46. English, Spanish. PMID 10089786
- [Background] Mate-Jimenez J, Munoz S, Vicent D, Pajares JM. Incidence and prevalence of ulcerative colitis and Crohn's disease in urban and rural areas of Spain from 1981 to 1988. J Clin Gastroenterol. 1994 Jan;18(1):27-31. doi: 10.1097/00004836-199401000-00008. PMID 8113581
- [Background] Sola Lamoglia R, Garcia-Puges AM, Mones Xiol J, Badosa Gallart C, Badosa Gallart J, Casellas F, Pujol Pi J, Varea V. [Chronic inflammatory intestinal disease in Catalonia (Barcelona and Gerona)]. Rev Esp Enferm Dig. 1992 Jan;81(1):7-14. Spanish. PMID 1547040
- [Background] Alonso P, Ulla M, Soriano M, Aquise M, Del Villar V. [Intestinal inflammatory disease in the province of Soria. Retrospective clinical and epidemiologic study from 1981 to 1990]. Rev Esp Enferm Dig. 1992 Aug;82(2):87-91. Spanish. PMID 1389554
- [Background] Brullet E, Rue M, Montserrat A, Gil M, Malet A, Mas P, Bonfill X. [A descriptive epidemiological study of ulcerative colitis in a community hospital (1985-1989)]. Med Clin (Barc). 1991 Jun 8;97(2):45-9. Spanish. PMID 1895781
- [Background] Hinojosa J, Primo J, Lledo S, Lopez A, Roig JV, Fernandez J. [Incidence of inflammatory bowel disease in Sagunto]. Rev Esp Enferm Dig. 1990 Nov;78(5):283-7. Spanish. PMID 2090171
- [Background] Ruiz V. Crohn's disease in Galicia, Spain. Scand J Gastroenterol Suppl. 1989;170:29-31; discussion 50-5. doi: 10.3109/00365528909091346. PMID 2617188
- [Background] Ruiz Ochoa V. [Epidemiologic study of Crohn's disease in Galicia from 1976 to 1983]. Rev Esp Enferm Apar Dig. 1984 Oct;66(4):273-9. No abstract available. Spanish. PMID 6515083
- [Background] Martinez G, Fernandez Y, Rodrigo Saez L, Martinez E. [Epidemiologic study of Crohn's disease in the Asturian region]. Rev Esp Enferm Apar Dig. 1983 Jun;63(6):534-41. No abstract available. Spanish. PMID 6878842
- [Background] Niewiadomski O, Studd C, Hair C, Wilson J, McNeill J, Knight R, Prewett E, Dabkowski P, Dowling D, Alexander S, Allen B, Tacey M, Connell W, Desmond P, Bell S. Health Care Cost Analysis in a Population-based Inception Cohort of Inflammatory Bowel Disease Patients in the First Year of Diagnosis. J Crohns Colitis. 2015 Nov;9(11):988-96. doi: 10.1093/ecco-jcc/jjv117. Epub 2015 Jun 30. PMID 26129692
- [Background] Bewtra M, Su C, Lewis JD. Trends in hospitalization rates for inflammatory bowel disease in the United States. Clin Gastroenterol Hepatol. 2007 May;5(5):597-601. doi: 10.1016/j.cgh.2007.01.015. Epub 2007 Mar 26. PMID 17382602
- [Background] Colombel JF, Sandborn WJ, Reinisch W, Mantzaris GJ, Kornbluth A, Rachmilewitz D, Lichtiger S, D'Haens G, Diamond RH, Broussard DL, Tang KL, van der Woude CJ, Rutgeerts P; SONIC Study Group. Infliximab, azathioprine, or combination therapy for Crohn's disease. N Engl J Med. 2010 Apr 15;362(15):1383-95. doi: 10.1056/NEJMoa0904492. PMID 20393175
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Reinisch W, Sandborn WJ, Hommes DW, D'Haens G, Hanauer S, Schreiber S, Panaccione R, Fedorak RN, Tighe MB, Huang B, Kampman W, Lazar A, Thakkar R. Adalimumab for induction of clinical remission in moderately to severely active ulcerative colitis: results of a randomised controlled trial. Gut. 2011 Jun;60(6):780-7. doi: 10.1136/gut.2010.221127. Epub 2011 Jan 5. PMID 21209123
- [Background] Sandborn WJ, Feagan BG, Rutgeerts P, Hanauer S, Colombel JF, Sands BE, Lukas M, Fedorak RN, Lee S, Bressler B, Fox I, Rosario M, Sankoh S, Xu J, Stephens K, Milch C, Parikh A; GEMINI 2 Study Group. Vedolizumab as induction and maintenance therapy for Crohn's disease. N Engl J Med. 2013 Aug 22;369(8):711-21. doi: 10.1056/NEJMoa1215739. PMID 23964933
- [Background] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, Van Assche G, Axler J, Kim HJ, Danese S, Fox I, Milch C, Sankoh S, Wyant T, Xu J, Parikh A; GEMINI 1 Study Group. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013 Aug 22;369(8):699-710. doi: 10.1056/NEJMoa1215734. PMID 23964932
- [Background] Fiocchi C. Integrating omics: the future of IBD? Dig Dis. 2014;32 Suppl 1:96-102. doi: 10.1159/000367836. Epub 2014 Dec 17. PMID 25531360
- [Background] Roda G, Caponi A, Benevento M, Nanni P, Mezzanotte L, Belluzzi A, Mayer L, Roda A. New proteomic approaches for biomarker discovery in inflammatory bowel disease. Inflamm Bowel Dis. 2010 Jul;16(7):1239-46. doi: 10.1002/ibd.21212. PMID 20127998
- [Background] Barcelo-Batllori S, Andre M, Servis C, Levy N, Takikawa O, Michetti P, Reymond M, Felley-Bosco E. Proteomic analysis of cytokine induced proteins in human intestinal epithelial cells: implications for inflammatory bowel diseases. Proteomics. 2002 May;2(5):551-60. doi: 10.1002/1615-9861(200205)2:53.0.CO;2-O. PMID 11987129
- [Background] Hardwidge PR, Rodriguez-Escudero I, Goode D, Donohoe S, Eng J, Goodlett DR, Aebersold R, Finlay BB. Proteomic analysis of the intestinal epithelial cell response to enteropathogenic Escherichia coli. J Biol Chem. 2004 May 7;279(19):20127-36. doi: 10.1074/jbc.M401228200. Epub 2004 Feb 26. PMID 14988394
- [Background] Hsieh SY, Shih TC, Yeh CY, Lin CJ, Chou YY, Lee YS. Comparative proteomic studies on the pathogenesis of human ulcerative colitis. Proteomics. 2006 Oct;6(19):5322-31. doi: 10.1002/pmic.200500541. PMID 16947118
- [Background] Shkoda A, Werner T, Daniel H, Gunckel M, Rogler G, Haller D. Differential protein expression profile in the intestinal epithelium from patients with inflammatory bowel disease. J Proteome Res. 2007 Mar;6(3):1114-25. doi: 10.1021/pr060433m. PMID 17330946
- [Background] Meuwis MA, Fillet M, Geurts P, de Seny D, Lutteri L, Chapelle JP, Bours V, Wehenkel L, Belaiche J, Malaise M, Louis E, Merville MP. Biomarker discovery for inflammatory bowel disease, using proteomic serum profiling. Biochem Pharmacol. 2007 May 1;73(9):1422-33. doi: 10.1016/j.bcp.2006.12.019. Epub 2006 Dec 20. PMID 17258689
- [Background] Nanni P, Parisi D, Roda G, Casale M, Belluzzi A, Roda E, Mayer L, Roda A. Serum protein profiling in patients with inflammatory bowel diseases using selective solid-phase bulk extraction, matrix-assisted laser desorption/ionization time-of-flight mass spectrometry and chemometric data analysis. Rapid Commun Mass Spectrom. 2007;21(24):4142-8. doi: 10.1002/rcm.3323. PMID 18022963
- [Background] Nanni P, Mezzanotte L, Roda G, Caponi A, Levander F, James P, Roda A. Differential proteomic analysis of HT29 Cl.16E and intestinal epithelial cells by LC ESI/QTOF mass spectrometry. J Proteomics. 2009 Jul 21;72(5):865-73. doi: 10.1016/j.jprot.2008.12.010. Epub 2009 Jan 8. PMID 19168159
- [Background] Hatsugai M, Kurokawa MS, Kouro T, Nagai K, Arito M, Masuko K, Suematsu N, Okamoto K, Itoh F, Kato T. Protein profiles of peripheral blood mononuclear cells are useful for differential diagnosis of ulcerative colitis and Crohn's disease. J Gastroenterol. 2010 May;45(5):488-500. doi: 10.1007/s00535-009-0183-y. Epub 2010 Jan 5. PMID 20049485
- [Background] M'Koma AE, Seeley EH, Washington MK, Schwartz DA, Muldoon RL, Herline AJ, Wise PE, Caprioli RM. Proteomic profiling of mucosal and submucosal colonic tissues yields protein signatures that differentiate the inflammatory colitides. Inflamm Bowel Dis. 2011 Apr;17(4):875-83. doi: 10.1002/ibd.21442. Epub 2010 Aug 30. PMID 20806340
- [Background] Presley LL, Ye J, Li X, Leblanc J, Zhang Z, Ruegger PM, Allard J, McGovern D, Ippoliti A, Roth B, Cui X, Jeske DR, Elashoff D, Goodglick L, Braun J, Borneman J. Host-microbe relationships in inflammatory bowel disease detected by bacterial and metaproteomic analysis of the mucosal-luminal interface. Inflamm Bowel Dis. 2012 Mar;18(3):409-17. doi: 10.1002/ibd.21793. Epub 2011 Jun 22. PMID 21698720
- [Background] Han NY, Choi W, Park JM, Kim EH, Lee H, Hahm KB. Label-free quantification for discovering novel biomarkers in the diagnosis and assessment of disease activity in inflammatory bowel disease. J Dig Dis. 2013 Apr;14(4):166-74. doi: 10.1111/1751-2980.12035. PMID 23320753
- [Background] Seeley EH, Washington MK, Caprioli RM, M'Koma AE. Proteomic patterns of colonic mucosal tissues delineate Crohn's colitis and ulcerative colitis. Proteomics Clin Appl. 2013 Aug;7(7-8):541-9. doi: 10.1002/prca.201200107. Epub 2013 May 8. PMID 23382084
- [Background] Townsend P, Zhang Q, Shapiro J, Webb-Robertson BJ, Bramer L, Schepmoes AA, Weitz KK, Mallette M, Moniz H, Bright R, Merrick M, Shah SA, Sands BE, Leleiko N. Serum Proteome Profiles in Stricturing Crohn's Disease: A Pilot Study. Inflamm Bowel Dis. 2015 Aug;21(8):1935-41. doi: 10.1097/MIB.0000000000000445. PMID 26199992
- [Background] Colombo M, Raposo G, Thery C. Biogenesis, secretion, and intercellular interactions of exosomes and other extracellular vesicles. Annu Rev Cell Dev Biol. 2014;30:255-89. doi: 10.1146/annurev-cellbio-101512-122326. Epub 2014 Aug 21. PMID 25288114
- [Background] Lugini L, Cecchetti S, Huber V, Luciani F, Macchia G, Spadaro F, Paris L, Abalsamo L, Colone M, Molinari A, Podo F, Rivoltini L, Ramoni C, Fais S. Immune surveillance properties of human NK cell-derived exosomes. J Immunol. 2012 Sep 15;189(6):2833-42. doi: 10.4049/jimmunol.1101988. Epub 2012 Aug 17. PMID 22904309
- [Background] Tran TH, Mattheolabakis G, Aldawsari H, Amiji M. Exosomes as nanocarriers for immunotherapy of cancer and inflammatory diseases. Clin Immunol. 2015 Sep;160(1):46-58. doi: 10.1016/j.clim.2015.03.021. Epub 2015 Apr 2. PMID 25842185
- [Background] Peche H, Heslan M, Usal C, Amigorena S, Cuturi MC. Presentation of donor major histocompatibility complex antigens by bone marrow dendritic cell-derived exosomes modulates allograft rejection. Transplantation. 2003 Nov 27;76(10):1503-10. doi: 10.1097/01.TP.0000092494.75313.38. PMID 14657694
- [Background] Mallegol J, van Niel G, Heyman M. Phenotypic and functional characterization of intestinal epithelial exosomes. Blood Cells Mol Dis. 2005 Jul-Aug;35(1):11-6. doi: 10.1016/j.bcmd.2005.04.001. PMID 15893486
- [Background] Zitvogel L, Regnault A, Lozier A, Wolfers J, Flament C, Tenza D, Ricciardi-Castagnoli P, Raposo G, Amigorena S. Eradication of established murine tumors using a novel cell-free vaccine: dendritic cell-derived exosomes. Nat Med. 1998 May;4(5):594-600. doi: 10.1038/nm0598-594. PMID 9585234
- [Background] Burisch J, Pedersen N, Cukovic-Cavka S, Brinar M, Kaimakliotis I, Duricova D, Shonova O, Vind I, Avnstrom S, Thorsgaard N, Andersen V, Krabbe S, Dahlerup JF, Salupere R, Nielsen KR, Olsen J, Manninen P, Collin P, Tsianos EV, Katsanos KH, Ladefoged K, Lakatos L, Bjornsson E, Ragnarsson G, Bailey Y, Odes S, Schwartz D, Martinato M, Lupinacci G, Milla M, De Padova A, D'Inca R, Beltrami M, Kupcinskas L, Kiudelis G, Turcan S, Tighineanu O, Mihu I, Magro F, Barros LF, Goldis A, Lazar D, Belousova E, Nikulina I, Hernandez V, Martinez-Ares D, Almer S, Zhulina Y, Halfvarson J, Arebi N, Sebastian S, Lakatos PL, Langholz E, Munkholm P; EpiCom-group. East-West gradient in the incidence of inflammatory bowel disease in Europe: the ECCO-EpiCom inception cohort. Gut. 2014 Apr;63(4):588-97. doi: 10.1136/gutjnl-2013-304636. Epub 2013 Apr 20. PMID 23604131
- [Background] Wisniewski JR, Zougman A, Nagaraj N, Mann M. Universal sample preparation method for proteome analysis. Nat Methods. 2009 May;6(5):359-62. doi: 10.1038/nmeth.1322. Epub 2009 Apr 19. PMID 19377485
- [Background] Gomez-Sanchez JA, Carty L, Iruarrizaga-Lejarreta M, Palomo-Irigoyen M, Varela-Rey M, Griffith M, Hantke J, Macias-Camara N, Azkargorta M, Aurrekoetxea I, De Juan VG, Jefferies HB, Aspichueta P, Elortza F, Aransay AM, Martinez-Chantar ML, Baas F, Mato JM, Mirsky R, Woodhoo A, Jessen KR. Schwann cell autophagy, myelinophagy, initiates myelin clearance from injured nerves. J Cell Biol. 2015 Jul 6;210(1):153-68. doi: 10.1083/jcb.201503019. PMID 26150392